CLINICAL TRIAL: NCT07396701
Title: Chinese Adaptive Randomised Pneumonia Trial With Respiratory Failure
Acronym: CARP-RF
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Hospital of Traditional Chinese Medicine (Other); Beijing Chest Hospital (Other); Shanghai University of Traditional Chinese Medicine (Other); Tianjin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZD01903003
Record Dates: First submitted 2025-11-23; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Severe Pneumonia With Respiratory Failure
MeSH Terms: interventions — Head-Down Tilt

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Receiving standard care alone (No Intervention): Receiving standard care alone
- Trendelenburg Position Group (Active Comparator): Trendelenburg Position: Standard care plus maintenance in the Trendelenburg position at -10° for ≥12 hours daily, continuing until sedation is discontinued and the patient regains consciousness (RASS 0).
  Interventions: Behavioral: Trendelenburg Position
- Traditional Chinese Medicine Formulation (Active Comparator): Traditional Chinese Medicine: Standard care plus a complementary TCM strategy prescribed by a licensed TCM practitioner. This includes the use of a tailored herbal formulation (Monarch:Trichosanthes 60g, Rhubarb 15g; Minister: Gypsum 30g, Bitter Apricot Seed 10g, Descurainia Seed 30g, Verbena 60g; Assistant: Glehnia 30g, Adenophora 30g, Astragalus 30g, Ophiopogon 15g, Schisandra 6g; Guide: Licorice 10g) One dose twice daily via oral/enteral route for 7 days.
  Interventions: Drug: Traditional Chinese Medicine Formulation

INTERVENTIONS:
Behavioral: Trendelenburg Position — Trendelenburg Position: Standard care plus Trendelenburg Position at -10° for ≥12 hours daily until sedation is discontinued and consciousness is recovered (RASS 0).
  Arms: Trendelenburg Position Group
Drug: Traditional Chinese Medicine Formulation — Traditional Chinese Medicine: Standard care plus a complementary TCM strategy prescribed by a licensed TCM practitioner. This includes the use of a tailored herbal formulation (Monarch:Trichosanthes 60g, Rhubarb 15g; Minister: Gypsum 30g, Bitter Apricot Seed 10g, Descurainia Seed 30g, Verbena 60g; Assistant: Glehnia 30g, Adenophora 30g, Astragalus 30g, Ophiopogon 15g, Schisandra 6g; Guide: Licorice 10g) One dose twice daily via oral/enteral route for 7 days.
  Arms: Traditional Chinese Medicine Formulation

SUMMARY:
1. Background Severe pneumonia with respiratory failure carries a high mortality rate. Preliminary evidence suggests potential benefits for interventions such as Trendelenburg Position and certain herbal formulations used within an integrative treatment framework. However, robust evidence from large-scale trials is lacking. This study utilizes an innovative adaptive platform trial design embedded within a continuous cohort to efficiently evaluate the efficacy and safety of these adjunctive interventions combined with standard care, with the inherent flexibility to incorporate future promising therapies.
2. Objectives Primary Objective: To evaluate whether adjunctive treatment with either Trendelenburg Position or Traditional Chinese Medicine (TCM) formulation, compared to standard care alone, reduces all-cause mortality at 28 days in patients with severe pneumonia and respiratory failure.

   Secondary Objectives: To assess the effects on clinical outcomes including incidence of ventilator-associated pneumonia (VAP), ventilator-free days, duration of mechanical ventilation and ICU stay, Sequential Organ Failure Assessment (SOFA) score trajectory, and oxygenation. To evaluate the safety profile of the interventions.
3. Study Design CARP-RF is a Chinese adaptive, randomised trial enrolling patients with pneumonia and respiratory failure. A continuously enrolled master cohort of eligible patients will be established. Within this cohort, eligible consenting participants will be centrally randomized in an unbalanced ratio of (1.5:1:1) to one of three parallel groups.
4. Participant Population Inclusion Criteria: Adult patients (≥18 years) admitted to the ICU, diagnosed with severe pneumonia per IDSA/ATS criteria (requiring invasive mechanical ventilation or meeting other major/minor criteria), under invasive mechanical ventilation and sedation (Richmond Agitation-Sedation Scale ≤ -1).

   Exclusion Criteria: Pregnancy, terminal illness, significant pulmonary fibrosis or lung cancer, known/suspected intracranial hypertension, increased intraocular pressure or recent eye surgery, and severe refractory hemodynamic instability.
5. Interventions All participants receive guideline-directed standard care for severe pneumonia. Control Group: Standard care only. Intervention Group 1: Standard care plus Trendelenburg Position at -10° for ≥12 hours daily until sedation is discontinued and consciousness is recovered (RASS 0).

   Intervention Group 2 (TCM): Standard care plus a complementary TCM strategy prescribed by a licensed TCM practitioner. This includes the use of a tailored herbal formulation (Monarch:Trichosanthes 60g, Rhubarb 15g; Minister: Gypsum 30g, Bitter Apricot Seed 10g, Descurainia Seed 30g, Verbena 60g; Assistant: Glehnia 30g, Adenophora 30g, Astragalus 30g, Ophiopogon 15g, Schisandra 6g; Guide: Licorice 10g). One dose twice daily via oral/enteral route for 7 days.
6. Outcome Measures Primary Outcome: All-cause mortality at 28 days after randomization. Key Secondary Outcomes: VAP incidence; Ventilator-free days at 28 days; duration of invasive mechanical ventilation; ICU and hospital length of stay; change in PaO₂/FiO₂ ratio; change in SOFA score.
7. Sample Size Approximately 1500 participants will be enrolled from multiple tertiary hospitals in China, accounting for consent rates, eligibility within the cohort, and a 5% attrition rate. The sample provides 80% power (alpha=0.05, two-sided) to detect an absolute mortality reduction from 30% to 20%.
8. Randomization, Blinding, and Consent Randomization is performed centrally via an Interactive Web Response System (IWRS), stratified by site and baseline SOFA score. The trial is open-label for caregivers and participants. Outcome assessors and data analysts will be blinded to treatment allocation. A two-stage consent process is used: broad consent for cohort data collection, followed by specific consent for the randomized intervention only for those allocated to an intervention group.
9. Data and Safety Monitoring An independent Data and Safety Monitoring Board (DSMB) will periodically review unblinded safety and efficacy data. Serious adverse events will be monitored and reported according to regulatory requirements. The DSMB may recommend protocol modifications, including early stopping for efficacy/futility or incorporation of new interventions into the adaptive platform.
10. Statistical Analysis The primary analysis will follow the intention-to-treat principle. Given the pragmatic design, a Compiler Average Causal Effect (CACE) analysis will supplement the primary analysis to estimate the effect among participants who adhere to the protocol. Pre-specified subgroup analyses will be conducted.
11. Ethical Considerations The protocol will be approved by the Institutional Review Board of the leading center and all participating sites. The study will be conducted in accordance with the Declaration of Helsinki and Good Clinical Practice guidelines.

ELIGIBILITY:
Inclusion Criteria: Adult patients (≥18 years) admitted to the ICU, diagnosed with severe pneumonia per IDSA/ATS criteria (requiring invasive mechanical ventilation or meeting other major/minor criteria), under invasive mechanical ventilation and sedation (Richmond Agitation-Sedation Scale ≤ -1).

Exclusion Criteria:

* Pregnancy, terminal illness
* Significant pulmonary fibrosis or lung cancer
* Known/suspected intracranial hypertension
* Increased intraocular pressure or recent eye surgery
* Spinal injury
* Severe refractory hemodynamic instability.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day mortality rate | 28day
  28-day mortality rate

SECONDARY OUTCOMES:
Incidence of Ventilator-Associated Pneumonia (VAP) | 28days
  Incidence of Ventilator-Associated Pneumonia (VAP)
Ventilator-free days (VFDs) within day 28 | 28days
  Ventilator-free days (VFDs) within day 28
Duration of mechanical ventilation (invasive or non-invasive), days | 28days
  Duration of mechanical ventilation (invasive or non-invasive), days
Length of Intensive Care Unit (ICU) stay, days | 28days
  Length of Intensive Care Unit (ICU) stay, days
Change in Sequential Organ Failure Assessment (SOFA) score | 28days
  The Sequential Organ Failure Assessment (SOFA) score is a validated tool used to quantify the degree of organ dysfunction in critically ill patients. It assesses six organ systems, each scored from 0 (normal) to 4 (most severe), with a total possible score of 0 to 24. A higher score indicates more severe organ failure.
  The components are:
  1. Respiratory System: Based on the PaO₂/FiO₂ ratio (mmHg).
  2. Coagulation: Based on platelet count (×10³/µL).
  3. Liver: Based on bilirubin level (mg/dL or µmol/L).
  4. Cardiovascular System: Based on mean arterial pressure (MAP) or the dose of required vasopressor/inotrope support.
  5. Central Nervous System: Based on the Glasgow Coma Scale (GCS) score.
  6. Renal System: Based on creatinine level (mg/dL or µmol/L) or urine output.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu TW, Zhang SW, Jiang H, Yang SW, Guo YJ, Ding MY, Li XC, Xu J, Lu HT, Ye HR, Hu YH, Li R, Wei YM, Song MF, Wang S, Zhang J, Feng QS, Xu XL. Effectiveness of Xuanbai Shengmai Decoction, a compound Chinese herbal medicine, on disease progress and viral RNA shedding in COVID-19 patients: A retrospective study of medical chart in China. J Integr Med. 2026 Jan;24(1):115-124. doi: 10.1016/j.joim.2025.10.001. Epub 2025 Oct 13. PMID 41177681
- [Background] Choi YS, Bang SO, Shim JK, Chung KY, Kwak YL, Hong YW. Effects of head-down tilt on intrapulmonary shunt fraction and oxygenation during one-lung ventilation in the lateral decubitus position. J Thorac Cardiovasc Surg. 2007 Sep;134(3):613-8. doi: 10.1016/j.jtcvs.2007.05.018. PMID 17723807
- [Background] Alsharifi A, Carter N, Irampaye A, Stevens C, Mejia E, Steier J, Rafferty GF. Ventilatory response to head-down-tilt in healthy human subjects. Exp Physiol. 2024 Dec;109(12):2134-2146. doi: 10.1113/EP092014. Epub 2024 Oct 24. PMID 39447579
- [Background] Li Bassi G, Panigada M, Ranzani OT, Zanella A, Berra L, Cressoni M, Parrini V, Kandil H, Salati G, Selvaggi P, Amatu A, Sanz-Moncosi M, Biagioni E, Tagliaferri F, Furia M, Mercurio G, Costa A, Manca T, Lindau S, Babel J, Cavana M, Chiurazzi C, Marti JD, Consonni D, Gattinoni L, Pesenti A, Wiener-Kronish J, Bruschi C, Ballotta A, Salsi P, Livigni S, Iotti G, Fernandez J, Girardis M, Barbagallo M, Moise G, Antonelli M, Caspani ML, Vezzani A, Meybohm P, Gasparovic V, Geat E, Amato M, Niederman M, Kolobow T, Torres A; Gravity-VAP Network. Randomized, multicenter trial of lateral Trendelenburg versus semirecumbent body position for the prevention of ventilator-associated pneumonia. Intensive Care Med. 2017 Nov;43(11):1572-1584. doi: 10.1007/s00134-017-4858-1. Epub 2017 Jun 20. PMID 29149418
- [Background] Kodamanchili S, Saigal S, Anand A, Panda R, Priyanka TN, Balakrishnan GT, Bhardwaj K, Shrivatsav P. Trendelenburg Ventilation in Patients of Acute Respiratory Distress Syndrome with Poor Lung Compliance and Diaphragmatic Dysfunction. Indian J Crit Care Med. 2022 Mar;26(3):319-321. doi: 10.5005/jp-journals-10071-24127. PMID 35519934